CLINICAL TRIAL: NCT02574572
Title: Evaluation of the Safety and Potential Effectiveness of Autologous Mesenchymal Stem Cells Transplantation in Subjects With Cervical Chronic and Complete Spinal Cord Injury
Brief Title: Autologous Mesenchymal Stem Cells Transplantation in Cervical Chronic and Complete Spinal Cord Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sao Rafael (Other)
Responsible Party: Principal Investigator, Ricardo Ribeiro dos Santos, PhD, Hospital Sao Rafael
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI-003
Record Dates: First submitted 2015-04-10; First posted 2015-10-14 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; Mesenchymal cells; Stem cells
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): Patients with spinal cord injury that will undergo laminectomy and autologous mesenchymal cells intralesional injection
  Interventions: Biological: Autologous mesenchymal cells transplantation

INTERVENTIONS:
Biological: Autologous mesenchymal cells transplantation — All patients will undergo laminectomy and autologous mesenchymal cells injection into the lesion area.

SUMMARY:
The purpose of this study is to analyze the safety and efficacy of autologous bone marrow mesenchymal stem cell transplantation in patients with cervical chronic and complete spinal cord injury.

DETAILED DESCRIPTION:
This is a pilot, phase I study, in a prospective cohort. The study population will consist of 10 patients who had spinal cord injury for at least 12 months, with cervical chronic and complete spinal cord injury, ASIA grade A.

A practitioner, a surgeon and a nurse will review the medical records of the patients to determine the presence / absence of inclusion / exclusion criteria. If the patient is a potential candidate for the study, an interview will be scheduled to review and confirm his/her eligibility.

Patients will undergo a series of clinical and neurological assessments and will also be submitted to the following procedures:

* Cell blood count;
* Biochemical analysis (measurement of electrolytes - sodium, potassium, magnesium);
* Renal function tests (urea and creatinine);
* Liver function tests;
* Coagulation profile;
* Metabolic profile (glucose, total cholesterol and fractions);
* Urine summary and culture;
* Serology required for blood transfusion and marrow transplant in Brazil;
* Electrocardiogram;
* Chest X-Ray;
* Bone densitometry;
* Urodynamic studies;
* Somatosensory evoked potential;
* Computed tomography of thoracic and lumbar spine;
* Magnetic resonance imaging of the thoracic and lumbar spine.

Also as part of the preoperative evaluation, the patients will respond to questions from the SF (Short Form) -36 questionnaire (for assessment of quality of life) and the questionnaires for the assessment of neuropathic pain.

Clinical follow-up will be kept for patients who suspend their participation in the study for any adverse event and / or laboratory abnormality, or for the patient's own desire, following insurance protocols. In addition to the clinical and surgical follow-up, specific medical care will be offered to patients who experience adverse events, until stabilization of the patient, even if the target date for completion of the study has been exceeded.

The candidates included in the study will be asked to voluntarily participate and give their informed written consent.

ELIGIBILITY:
Inclusion Criteria:

* Blunt spinal cord injury at cervical level, between C5 and C7, or penetrating spinal cord injury, at the same level, provided that the mechanism of injury had been spinal shock, ischemia or hematoma, with at least 12 months of injury;
* ASIA grade A;
* Signing of the written consent.

Exclusion Criteria:

* Spinal cord injuries by sharp objects, firearms, and not traumatic or congenital causes, even if at different levels of the spinal cord;
* Concomitant brain injuries;
* Diabetes mellitus type 1 or 2 as defined by fasting glucose above 126 mg / use of medication and medical history;
* Infectious processes in acute and / or chronic course, confirmed by additional tests and / or medical history;
* Immunodeficiency, autoimmune diseases and neoplastic processes, confirmed by additional tests and / or medical history;
* Terminal, neurodegenerative, primary hematologic and musculoskeletal diseases confirmed by additional tests and / or past medical history;
* Osteopathies reflecting increased risk for bone marrow puncture;
* Coagulopathies;
* Severe organ failure (heart, kidney or liver), confirmed by additional tests or medical history;
* Pregnancy or lactation;
* Clinical complications that hinder or contraindicate the surgical procedure;
* Use of metallic implants near vascular structures (such as cardiac pacemaker), or other contraindication to magnetic resonance imaging;
* Psychiatric disorders, psychosocial and cognitive impairment confirmed by medical evaluation;
* Abusive use of alcohol and / or illegal substances use;
* Participation in other clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by magnetic resonance imaging | 12 months

SECONDARY OUTCOMES:
Functional improvement in ASIA (American Spinal Injury Association) grade | 12 months
  The investigators will evaluate the conversion rate from ASIA A to B or C in 12 months.
Functional improvement regarding the AIS (ASIA Impairment Scale) scores (light touch, pin prik and motor force) | 12 months
  AIS (ASIA Improvement Scale) degree on the ASIA score will be assessed in order to evaluate sensitivity and motor force in 12 months.
Improvements in sensorial mapping and neuropathic pain | 12 months
  The patients will be submitted to specific questionnaires and clinical examinations in order to evaluate improvements in sensorial mapping and neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Ribeiro-dos-Santos, PhD, Principal Investigator — Hospital São Rafael; Milena BP Soares, PhD, Study Director — Hospital São Rafael; Bruno SF de Souza, MD, Msc, Study Chair — Hospital São Rafael; Ticiana F Larocca, MD, Msc, Study Chair — Hospital São Rafael; Rodrigo L Alves, MD, PhD, Study Chair — Hospital São Rafael; Carolina T Macedo, MD, MSc, Study Chair — Hospital São Rafael; André C Matos, MD, Study Chair — Hospital São Rafael; Cristiane F Villarreal, PhD, Study Chair — Fundação Oswaldo Cruz; Antônio Olímpio S Moura, MD, Study Chair — Hospital São Rafael; Eduardo Brazão, MD, Study Chair — Hospital São Rafael; Kátia N Silva, MSc, Study Chair — Hospital São Rafael; Daniela N Silva, MSc, Study Chair — Hospital São Rafael; Clarissa LM de Souza, MD, Study Chair — Hospital São Rafael
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Macedo CT, de Freitas Souza BS, Villarreal CF, Silva DN, da Silva KN, de Souza CLEM, da Silva Paixao D, da Rocha Bezerra M, da Silva Moura Costa AO, Brazao ES, Marins Filho JP, Matos AC, Dos Santos RR, Soares MBP. Transplantation of autologous mesenchymal stromal cells in complete cervical spinal cord injury: a pilot study. Front Med (Lausanne). 2024 Sep 12;11:1451297. doi: 10.3389/fmed.2024.1451297. eCollection 2024. PMID 39328312